CLINICAL TRIAL: NCT06369688
Title: Effect of IDEAL SKIIN CARES Bundle to Prevent Hospital-acquired Pressure Injury: A Cluster Randomized Clinical Trial
Brief Title: IDEAL SKIIN CARES Bundle to Prevent Pressure Injury
Acronym: IdealSkinCares
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Tehran University of Medical Sciences (Other); Hamadan University of Medical Science (Other); Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Professor, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Baqiyatallah University
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pressure Ulcer; Pressure Injury; Bed Sore; Pressure Sore; Decubitus Sore; Decubitus Ulcer; Skin Ulcer
Keywords: Pressure Injury; Care Bundle; Hospital-acquired pressure injury; Randomized Clinical Trial; IDEAL SKIIN CARES
MeSH Terms: conditions — Pressure Ulcer; Skin Ulcer

STUDY DESIGN:
Intervention Model Description: C-RCT will be conducted with a three-arm parallel design and a 1:1:1 allocation ratio. The experimental groups will consist of two arms: the intervention group and the placebo group. The third arm will be the control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this placebo-controlled trial, patients will be blinded to their group allocations. Additionally, WSNs, who are trained for delivering special PIP care bundles, as well as nursing staff who are responsible for measuring wounds and collecting data, and data analyst, will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): Educational packages including a pamphlet, brochure, and visual poster that outlines three key components of the IDEAL SKIIN CARES bundle (Education, Assessment of patient's condition and Care intervention) will be provided along with sub-items. These materials will be explained in detail by a trained research assistant in a workshop. Patients will be encouraged by the research assistant to actively participate in PIP self-care activities following the IDEAL SKIIN CARES approach shortly after recruitment and will continue to provide patient education throughout the study period. This training will begin before data collection and will be maintained as needed. Each hospital's study investigator will oversee the training activities at their site to guarantee consistency and adherence to the intervention protocol. In addition, patients will receive the IDEAL SKIIN CARES bundle from WSNs.
  Interventions: Other: IDEAL SKIIN CARES bundles; Other: IDEAL SKIIN CARES bundles workshop
- Placebo group (Placebo Comparator): The placebo group will receive training in an unrelated topic, specifically respiratory care. This training will involve the distribution of educational pamphlets, brochures, and visual posters outlining key aspects of respiratory care, mirroring the approach taken with the intervention group. Despite the focus on respiratory care education, patients in the placebo group will also benefit from specialized PIP care through the IDEAL SKIIN CARES bundle, administered by trained WSNs. These WSNs will provide interventions focused on PIP strategies based on the IDEAL SKIIN CARES bundle, ensuring that patients in the placebo group receive comprehensive wound care support throughout the study period.
  Interventions: Other: IDEAL SKIIN CARES bundles; Other: Respiratory care workshop
- Control group (No Intervention): The control group will not receive any relevant or irrelevant training or educational materials. They will only receive routine standard care for the PIP care bundle, following the care plans as routine by the hospital.

INTERVENTIONS:
Other: IDEAL SKIIN CARES bundles — The investigators developed a specialized PIP care bundle, named IDEAL SKIIN CARES, through extensive review of literature and expert insights, which will be utilized for training WSNs and patients in the intervention group. This comprehensive bundle comprises 15 key components aimed at effectively preventing PIs: (1) Incontinence care status; (2) Dehydration status; (3) Elevate at-risk surfaces; (4) Attention to attached devices to skin; (5) Lotion use; (6) Skin assessment; (7) Keeping repositioning; (8) Individualized up-to-date knowledge; (9) Individualized medical devices selection; (10) Nutrition status; (11) Caregiver (formal and informal) participation; (12) Activity assessment; (13) Reducing friction/shear forces; (14) Evaluate hemodynamic instability; (15) and Scrutinizing comorbidities.
  Arms: Intervention group; Placebo group
Other: IDEAL SKIIN CARES bundles workshop — IDEAL SKIIN CARES bundles will be explained in detail by a trained research assistant in a workshop. This workshop is different from clinical training and following up about the IDEAL SKIIN CARES bundles.
  Arms: Intervention group
Other: Respiratory care workshop — An unrelated topic, specifically respiratory care will be held in a workshop. This training will involve the distribution of educational pamphlets, brochures, and visual posters outlining key aspects of respiratory care
  Arms: Placebo group

SUMMARY:
The study will be a multi-center, triple-blinded, cluster randomized controlled trial (c-RCT) conducted with a three-arm parallel design and a 1:1:1 allocation ratio. The experimental groups will consist of two arms: the intervention group, where patients will receive training in relevant pressure injury care bundles, and the placebo group, where patients will receive training in an irrelevant topic like respiratory care. Both intervention and placebo groups will receive specialized pressure injury prevention (PIP) care bundle from trained wound specialist nurses (WSNs). The third arm will be the control group comprising patients who do not undergo any training course and will receive only routine standard care for PIP care bundle. The aim of c-RCT will be to compare the incidence of hospital-acquired pressure injury (HAPI) in the three study groups and to provide detailed evidence on the effect of the developed pressure injury care bundle, administered by WSNs on the development of HAPI in trained hospitalized patients, as opposed to those receiving routine standard care for PIP care bundle without training.

DETAILED DESCRIPTION:
The investigators developed a specialized PIP care bundle, named IDEAL SKIIN CARES, through extensive review of literature and expert insights, which will be utilized for training WSNs and patients in intervention group. This comprehensive bundle comprises 15 key components aimed at effectively preventing PIs: (1) Incontinence care status; (2) Dehydration status; (3) Elevate at-risk surfaces; (4) Attention to attached devices to skin; (5) Lotion use; (6) Skin assessment; (7) Keeping repositioning; (8) Individualized up-to-date knowledge; (9) Individualized medical devices selection; (10) Nutrition status; (11) Caregiver (formal and informal) participation; (12) Activity assessment; (13) Reducing friction/shear forces; (14) Evaluate hemodynamic instability; (15) and Scrutinizing comorbidities. These components are categorized into three groups to facilitate understanding and enhance patient engagement in PIP care: (1) Education; (2) assessment of patient's condition; and (3) Care intervention. Therefore, the investigators will conduct a c-RCT with three arm parallel design for hospitalized patients to assessed the effect of IDEAL SKIIN CARES bundle to prevent of occurrence HAPI in three groups of study and compare with routine standard care for PIP care bundle.

ELIGIBILITY:
Inclusion Criteria:

* be adults aged 18 years or older;
* have been hospitalized for a minimum of 48 hours;
* be willing to participate.

Exclusion Criteria:

* patients with significant pre-existing skin conditions or injuries that make it difficult to observe skin integrity;
* have existing PIs or vascular ulcers upon admission to the hospital (pressure injuries defined by the National Pressure Ulcer Advisory Panel);
* be at risk of PIs due to limited mobility (requiring physical or mechanical assistance to reposition or move);
* individuals with urinary or fecal incontinence, mental illness, or severe cognitive impairment upon hospital admission;
* patients who are hospitalized in day-surgery, critical care, emergency, maternity, pediatrics, mental health and dialysis units;
* admitted to the hospital for >28 days;
* those with prior experience of PIs or training in PIs care and prevention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1620 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital-acquired pressure injury (HAPI) | Within 48 hours of hospital admission until they reach the trial endpoints of hospital discharge or 28 days
  All patients in the three groups will be closely monitored for the development of HAPI. Two independent and experienced WSNs will oversee the intervention and placebo groups, while two independent and experienced research assistants will supervise the control group. They will conduct separate examinations of the patients to assess the presence or absence of PI, following the NPUAP guidelines. These assessments will occur three times a day during morning, evening, and night shifts to ensure comprehensive monitoring of at-risk patients, and with daily evaluations for patients without PI risk factors. The occurrence time of PI will be recorded for each patient based on the day. To ensure consistency and accuracy in PI assessment, the agreement between the two assessors will be evaluated using the Kappa agreement test for inter-rater reliability

SECONDARY OUTCOMES:
Pressure Injury Stage | Within 48 hours of hospital admission until they reach the trial endpoints of hospital discharge or 28 days
  Wound specialist nurses and experienced research assistants will determine the stage of PIs among patients and monitor the progression of PI stages (increased severity in PI stages) in all three study groups. The stages of a pressure ulcer typically range from Stage 1 to Stage 4, with each stage indicating the severity of tissue damage. The assessment of PI stages will involve evaluating factors such as skin integrity, tissue involvement, and the presence of necrosis. Any changes in the stage of a PI will be carefully documented to track the progression of the injury over time. To ensure consistency and accuracy in PI stage determination, the agreement between the two assessors will be evaluated using the Kappa agreement test for inter-rater reliability on stage of PI.
Patient participation in care | Within 48 hours of hospital admission until they reach the trial endpoints of hospital discharge or 28 days
  When patients reach the trial endpoint, the assessor (the research assistants and WSNs) will utilize the Patient Participation Scale as a secondary outcome measure.
Healthcare costs | Within 48 hours of hospital admission until they reach the trial endpoints of hospital discharge or 28 days
  The costs linked to providing the IDEAL SKIIN CARES bundle, including time spent on patient education, training WSNs, and developing educational resources like brochures, posters, and pamphlets, will be gathered for all participants in the trial. Additionally, data on the length of hospital stays will be collected. Over a 28-day observational period, detailed micro-costing data will be collected by a dedicated research assistant. Specifically, the number of repositioning episodes per participant, the clinical staff required for repositioning, and the nurse time needed per repositioning will be determined. Other resources utilized for IDEAL SKIIN CARES or standard care bundles, such as special mattresses, skincare products, and incontinence care, will also be documented. The direct costs will then be allocated to each resource unit using established costing references.
Self-report Patient participation in care | Within 48 hours of hospital admission until they reach the trial endpoints of hospital discharge or 28 days
  Patients will be asked to self-report their level of participation in PIP by providing a score from 0 to 10. This self-assessment will offer insights into the patient's perception of their involvement in their care plan.

CONTACTS AND LOCATIONS:
Overall Officials: Amir vahedian-azimi, Professor, Principal Investigator — Baqiyatallah University of Medical Sciences, Tehran, Iran.; Keivan Goharimoghadam, Professor, Study Director — Tehran University of Medical Scienecs, Tehran, Iran; Farshid Rahimi-bashar, Professor, Study Director — Hamadan University of Medical Sciences, Hamadan, Iran.; Ata Mahmoodpoor, Professor, Study Director — Tabriz university of Medical Sciences, Tabriz, Iran.